CLINICAL TRIAL: NCT01385930
Title: A New Concept for Lifestyle Change, Dietary Advice on Prescription (DAP) in Combination With Motivational Interviewing (MI), Social Support and Mobile Services
Brief Title: Dietary Advice on Prescription in Kungsbacka
Acronym: DAP_K
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Halmstad University (Other)
Collaborators: Carema (Unknown); Region Halland (Other)
Responsible Party: Gunnar Johansson, professor, Halmstad University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Halm30118
Record Dates: First submitted 2011-06-29; First posted 2011-06-30 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-03

CONDITIONS: Overweight
Keywords: Overweight; Obesity; lifestyle counseling
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental): Lifestyle counseling
  Interventions: Behavioral: Lifestyle counseling
- Control group (No Intervention): Control group

INTERVENTIONS:
Behavioral: Lifestyle counseling — Lifestyle counseling
  Arms: Lifestyle counseling

SUMMARY:
The aim of the study is to evaluate self-reported adherence to and the effects of an intervention model consisting of individualized prescribed dietary advice (DAP) in combination with Motivational Interviewing (MI), social support and mobile services in obese patients in primary health care. The specific aim is to relate effects of the intervention model to self-reported health, biomarkers for coronary heart disease, diabetes, some cancer forms, sleep duration and quality, health economy, oral health, dietary intake and physical activity.

This is a two-armed randomized controlled study. The arms are: 1) Control group (care as usual) and 2) Experimental group (MoR). The volunteers will be consecutively, for each sex, randomized to the experimental and the control group, respectively.

The experimental group will receive DAP together with Motivational interviewing up to six months after the start of the study. From six months up to 24 months the participants will receive social support online and mobile services.

The control group will receive dietary information according to the "Habo model". The previously mentioned diet will be recommended to both the control group and the experimental group since it is the method in which the investigators give the information they want to study and not the diet per se. Thus, it is only the way the investigators give dietary information that differs between the groups.

The study also includes qualitative interviews. The aim of these studies is to gain understanding of patients' and health professionals' experience and attitudes around food, lifestyle and support functions associated with dietary change. The sampling approach involves the purposeful selection of cases with a wide range of variation, which means that the researcher selects people who are able to provide rich information about the current issue. To achieve diversity, it is useful that both women and men are involved in the studies, as well as people of different ages and with different experiences of providing or receiving dietary advice. About 15-20 people will participate in each interview study.

DETAILED DESCRIPTION:
The investigators assume a difference in BMI (body mass index; kg/m x m) of 2 units, a standard deviation of 4.5 units, a power of 80 %, an alfa error of 5 % I a two-tailed test, the investigators would need at least 80 individuals in the experimental group and in the control group, respectively.

With 80 individuals in each group and the assumption of 5 % adherence (4 individuals) in the control group, the investigators would be able to detect an adherence of 21 % or higher (at least 17 individuals) in the experimental group with 80 % power. The alfa error is set to 5 % in a two-tailed test with the null hypothesis that the adherence is the same in both groups.

Therefore the investigators plan a study with at least 100 individuals in each group and assume that 20 % will not complete the study.

The evaluation of the quantitative studies will be performed in three ways: 1) Process evaluation, that will focus on intermediate outcomes such as knowledge, attitudes, motivation and readiness for change. 2) Effect evaluation will be used to evaluate the effect of the intervention programme on the subjects' behavior such as dietary intake and physical activity level. 3) Outcome evaluation will measure the total effect of the intervention programme, in this case variables that measures indicators for health and disease, such as SF-36, EQ-5D, SHIS, serum cholesterol, blood pressure, BMI, waist circumference etc.

Intention-to-treat (ITT) analysis will be used to assess effects on outcome measures. Variables not normally distributed will be logarithmically transformed. Paired t-test will be used to assess change within groups and unpaired t-tests to compare mean changes between groups. Non-parametric statistics, Wilcoxon Signed Ranks Test and Mann-Whitney U-Test will be used for ordinal data such as questionnaires. Two-tailed tests will be used and a p-value less than 0.05 will be considered statistically significant.

Qualitative data will be analyzed by content analysis.

ELIGIBILITY:
Inclusion Criteria:

* BMI 28-35

Exclusion Criteria:

* Severe disease

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
BMI | two years
  Lifestyle intervention

SECONDARY OUTCOMES:
LDL cholesterol | two years
  Lifestyle intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Carema husläkarna, Kungsbacka, Halland County, Sweden